CLINICAL TRIAL: NCT05252728
Title: Altered Faecal Microbiome and Metabolome in Childhood-onset Type 1 Diabetes, Adult-onset Type 1 Diabetes and Type 2 Diabetes
Brief Title: Altered Faecal Microbiome and Metabolome in CT1D, AT1D and T2D
Status: Completed | Type: Observational
Sponsor: Second Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, Yang Xiao, Associate Professor, Department of Metabolism and Endocrinology, Institute of Metabolism and Endocrinology, National Clinical Research Center for Metabolic Diseases, Second Xiangya Hospital, Central South University, Second Xiangya Hospital of Central South University
Other Study IDs: 2021AT1DDC
Record Dates: First submitted 2022-02-13; First posted 2022-02-23 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-04

CONDITIONS: Type 1 Diabetes Mellitus Maturity Onset
Keywords: adult-onset type 1 diabetes; microbiota; metabolomics

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Feces，serum
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Healthy control
- Childhood-onset type 1 diabetes
- Adult-onset type 1 diabetes
- Type 2 diabetes

SUMMARY:
To elucidate the characteristics of global gut microbiota and fecal/serum metabolites in patients with childhood-onset type 1 diabetes, adult-onset type 1 diabetes or type 2 diabetes.

DETAILED DESCRIPTION:
Type 1 diabetes is caused by autoimmune destruction of pancreatic beta cells, leading to severe insulin deficiency and requiring insulin therapy. It is typically considered a disease of childhood and adolescence, but recent epidemiological data have shown that over half of all new-onset type 1 diabetes cases occur in adults worldwide. There are genetic, immune and metabolic differences between adult- and childhood-onset type 1 diabetes, revealing the underlying molecular basis of type 1 diabetes onset at diverse ages may differ. Accurate diagnosis is of great importance because the best treatment for different types of diabetes is divergent. Misdiagnosing type 2 diabetes as type 1 diabetes can lead to unnecessary initial insulin therapy, resulting in higher costs and more side effects. Thus, it is critical to identify the molecular basis and new diagnostic biomarkers for adult-onset type 1 diabetes.

Nonetheless, environmental exposures, in particular the immense intestinal microbiota and its derivatives, have been widely investigated. Indeed, patients with childhood-onset type 1 diabetes or type 2 diabetes exhibit compositional alterations in gut microbiota. However, gut microbiota in adult-onset type 1 diabetes has not been elucidated, and little is known about the shared and distinct microbial characteristics in adult-onset type 1 diabetes versus childhood-onset type 1 diabetes or type 2 diabetes.

Thus, this study is a cross-sectional study. 4 groups of subjects were recruited for metagenome and metabolome analysis, including healthy controls and patients with childhood-onset type 1 diabetes, adult-onset type 1 diabetes or type 2 diabetes. All subjects recruited meet the inclusion or exclusion criteria and written informed consent was obtained from each participant at enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. Diabetes diagnosed according to the report of WHO in 1999；
2. Aged between 5 and 70 years old;

Exclusion Criteria:

1. Severe chronic cardiovascular or cerebrovascular disease；
2. Severe abnormalities in liver or renal function;
3. Hyperthyroidism; or other autoimmune diseases;
4. Tumors, surgery or pregnancy;
5. Treatments with oral hypoglycemic agents or immunomodulators;
6. Subjects who had taken probiotics, prebiotics within one week or antibiotics within one month.

Ages: 5 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with childhood-onset type 1 diabetes, adult-onset type 1 diabetes or type 2 diabetes. Healthy conrols recruited at the Second Xiangya Hospital of Central South University in Changsha.
Sampling Method: Non-Probability Sample
Enrollment: 372 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Differences of β diversity of gut microbiota between diabetic groups and healthy control. | at baseline
  β diversity is based on metagenome analysis and statistical significance is estimated by permutational multivariate analysis of variance.

CONTACTS AND LOCATIONS:
Overall Officials: Yang Xiao, MD/PhD, Principal Investigator — Institute of Metabolism and Endocrinology, Second Xiangya Hospital, Central South University, China
Locations (1):
- Institute of Metabolism and Endocrinology, Second Xiangya Hospital, Central South University, Changsha, Hunan, China

REFERENCES:
- [Background] Holt RIG, DeVries JH, Hess-Fischl A, Hirsch IB, Kirkman MS, Klupa T, Ludwig B, Norgaard K, Pettus J, Renard E, Skyler JS, Snoek FJ, Weinstock RS, Peters AL. The Management of Type 1 Diabetes in Adults. A Consensus Report by the American Diabetes Association (ADA) and the European Association for the Study of Diabetes (EASD). Diabetes Care. 2021 Nov;44(11):2589-2625. doi: 10.2337/dci21-0043. Epub 2021 Sep 30. PMID 34593612
- [Background] Leslie RD, Evans-Molina C, Freund-Brown J, Buzzetti R, Dabelea D, Gillespie KM, Goland R, Jones AG, Kacher M, Phillips LS, Rolandsson O, Wardian JL, Dunne JL. Adult-Onset Type 1 Diabetes: Current Understanding and Challenges. Diabetes Care. 2021 Nov;44(11):2449-2456. doi: 10.2337/dc21-0770. PMID 34670785
- [Background] Fang Y, Zhang C, Shi H, Wei W, Shang J, Zheng R, Yu L, Wang P, Yang J, Deng X, Zhang Y, Tang S, Shi X, Liu Y, Yang H, Yuan Q, Zhai R, Yuan H. Characteristics of the Gut Microbiota and Metabolism in Patients With Latent Autoimmune Diabetes in Adults: A Case-Control Study. Diabetes Care. 2021 Dec;44(12):2738-2746. doi: 10.2337/dc20-2975. Epub 2021 Oct 7. PMID 34620611
- [Background] Honkanen J, Vuorela A, Muthas D, Orivuori L, Luopajarvi K, Tejesvi MVG, Lavrinienko A, Pirttila AM, Fogarty CL, Harkonen T, Ilonen J, Ruohtula T, Knip M, Koskimaki JJ, Vaarala O. Fungal Dysbiosis and Intestinal Inflammation in Children With Beta-Cell Autoimmunity. Front Immunol. 2020 Mar 19;11:468. doi: 10.3389/fimmu.2020.00468. eCollection 2020. PMID 32265922
- [Derived] Hu J, Ding J, Li X, Li J, Zheng T, Xie L, Li C, Tang Y, Guo K, Huang J, Liu S, Yan J, Peng W, Hou C, Wen L, Xu A, Zhou Z, Xiao Y. Distinct signatures of gut microbiota and metabolites in different types of diabetes: a population-based cross-sectional study. EClinicalMedicine. 2023 Aug 3;62:102132. doi: 10.1016/j.eclinm.2023.102132. eCollection 2023 Aug. PMID 37593224